CLINICAL TRIAL: NCT02125916
Title: Evaluating the Effect of Oxygentherapy on Concentration at Chronic Lung Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Driving simulation COLD & ILD
Record Dates: First submitted 2014-04-23; First posted 2014-04-29 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Lung Diseases, Interstitial; Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Lung Diseases, Interstitial; Pulmonary Disease, Chronic Obstructive | interventions — Oxygen

ARMS (4):
- COLD without long term oxygen therapy (Experimental): Driving in the simulator two times, one time with and one time without oxygen therapy
  Interventions: Other: oxygen therapy
- COLD with long term oxygen therapy (Experimental): Driving in the simulator two times, one time with and one time without oxygen therapy
  Interventions: Other: oxygen therapy
- ILD without long term oxygen therapy (Experimental): Driving in the simulator two times, one time with and one time without oxygen therapy
  Interventions: Other: oxygen therapy
- Controls (No Intervention): Driving in the simulator one time without oxygen therapy

INTERVENTIONS:
Other: oxygen therapy
  Arms: COLD with long term oxygen therapy; COLD without long term oxygen therapy; ILD without long term oxygen therapy

SUMMARY:
The objective is to study the cognitive functions in patients with chronic obstructive lung disease (COLD) and patients with interstitial lung disease (ILD) compared to healthy controls. The cognitive functions are tested with and without oxygen therapy to clarify the effect of oxygen therapy. Driving simulations is used to test the cognitive functions.

The hypothesis is that patients with chronic lung disease have decreased cognitive functions and that oxygen therapy will increase their cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

* COLD with forced expiratory volume at one second (FEV1) <50%, without long term oxygen therapy
* COLD with FEV1 <50%, with long term oxygen therapy
* ILD with diffusion capacity of lung for carbon monoxide (DLCO) < 50%, without long term oxygen therapy

Exclusion Criteria:

* comorbidity which decreases cognitive function
* comorbidity which decreases concentration
* physical comorbidity which makes it impossible to complete the test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-07; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Standard deviation from the centre of the road | During the 45 min. of driving in the simulator
  Measuring how far from the centre of the road the patient has been driving in the driving simulation
Number of nil responses | During the 45 min. of driving in the simulator
  Measuring the number of times the patients doesn't react to the number "2" on the screen
Response time | During the 45 min. of driving in the simulator
  Measuring the mean amount of response time from the number "2" appears on the screen until the patient reacts
Number of off-road events per hour | During the 45 min. of driving in the simulator
  The number of times the car is off-road during the driving simulation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Skovhus Prior, MD, Principal Investigator — Department of pulmonology and allergology, Aarhus University Hospital, NBG; Ole Hilberg, Dr.med, MD, Study Chair — Department of pulmonology and allergology, Aarhus University Hospital, NBG
Locations (1):
- Department of pulmonology and allergology, Aarhus University Hospital, NBG, Aarhus, Denmark

REFERENCES:
- [Derived] Skovhus Prior T, Troelsen T, Hilberg O. Driving performance in patients with chronic obstructive lung disease, interstitial lung disease and healthy controls: a crossover intervention study. BMJ Open Respir Res. 2015 Dec 17;2(1):e000092. doi: 10.1136/bmjresp-2015-000092. eCollection 2015. PMID 26719805